CLINICAL TRIAL: NCT05101187
Title: Phase III, Adjudicator-blinded, Randomised Study to Evaluate Efficacy and Safety of Treatment With Olorofim Versus Treatment With AmBisome® Followed by Standard of Care in Patients With Invasive Fungal Disease Caused by Aspergillus Species
Brief Title: Olorofim Aspergillus Infection Study
Acronym: OASIS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: F2G Biotech GmbH (Industry)
Collaborators: Iqvia Pty Ltd (Industry); Shionogi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F901318/0041
Record Dates: First submitted 2021-09-07; First posted 2021-11-01 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Invasive Aspergillosis
Keywords: Invasive fungal disease (IFD); Aspergillus species; Olorofim; Non-azole antifungal; Azole resistance
MeSH Terms: conditions — Invasive Fungal Infections | interventions — olorofim; liposomal amphotericin B

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Adjudicator and sponsor-blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Olorofim (Active Comparator): Olorofim versus AmBisome followed by Standard of Care (SOC)
  Interventions: Drug: Olorofim
- AmBisome (Active Comparator): Olorofim versus AmBisome followed by Standard of Care (SOC)
  Interventions: Drug: AmBisome®

INTERVENTIONS:
Drug: Olorofim — Loading Dose: 5 tablets (150 mg) to be taken twice daily at a 12-hour (± 1 hour) interval on Day 1 Maintenance Dose: 3 tablets (90 mg) to be taken twice daily at 12-hour (± 1 hour) intervals from Day 2 until Day 84 (± 7 days)
  Other Names: Olorofim (F901318)
  Arms: Olorofim
Drug: AmBisome® — Initial course of at least 10 days of AmBisome® administered daily at a dose of 3 mg/kg by IV infusion over a 30- to 60-minute period or according to local guidelines Administration of SOC will follow international, national, or local guidelines and product labelling.
  Other Names: AmBisome® (liposomal amphotericin B)
  Arms: AmBisome

SUMMARY:
The purpose of this study is to compare treatment with olorofim versus treatment with AmBisome® followed by standard of care (SOC) in patients with IFD caused by proven IA or probable lower respiratory tract disease Aspergillus species (invasive aspergillosis, IA).

DETAILED DESCRIPTION:
The mortality rate in immunosuppressed patients with IA is high even with effective modern antifungal drug treatment. Intrinsic and acquired resistance to azoles and amphotericin B, the two most effective classes of treatment, have been identified in Aspergillus species and are linked to this increased mortality.

Currently marketed antifungal drugs have limitations including limited dosage forms, DDIs, and significant adverse reactions.

For patients with IA who do not respond to or cannot tolerate a triazole therapy, treatment options are even more limited.

Olorofim is an antifungal candidate with a novel mechanism of action offering activity against resistant organisms, differences in safety profile, along with oral dosing, predictable and reliable pharmacokinetic (PK) profile and limited potential for DDIs.

The present study is designed to compare the efficacy, safety, and tolerability of olorofim with that of AmBisome® followed by guideline-based hierarchy standard of care (SOC) in patients with IA whose infection is either refractory to or unsuitable for azole therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients ages over 18 years and weighing more than 30 kg
2. Patients with proven IA at any site or probable LRTD IA per EORTC/MSG 2019 criteria as adapted for this study and where the duration of specific therapy for this episode of IA has been ≤ 28 days. For purposes of this inclusion, the duration of specific therapy includes any mould-active therapy given for this episode of IA whether subsequently judged potentially effective or not.
3. Patients requiring therapy with an antifungal agent other than a mould-active azole, and who have had ≤ 96 hours of potentially effective prior therapy. Potentially effective prior therapy includes any agent to which the infecting strain of Aspergillus is likely to be susceptible. There are no exclusions or limitations on such agents (eg, AmBisome® is permitted) other than their duration.
4. AmBisome® is an appropriate therapy for the patient.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding.
2. Known history of allergy, hypersensitivity, or any serious reaction to any component of the study drug
3. Patients with only chronic aspergillosis, aspergilloma, or allergic bronchopulmonary aspergillosis.
4. Suspected mucormycosis (zygomycosis).
5. Patients with a known active second fungal infection of any type, other than candidiasis that can be treated with fluconazole.
6. The requirement for ongoing use of echinocandin as Candida prophylaxis.
7. Microbiological findings (eg, bacteriological, virological) or other potential conditions that are temporally related and suggest a different aetiology for the clinical features.
8. Human immunodeficiency virus (HIV) infection but not currently receiving antiretroviral therapy.
9. Patients with a baseline prolongation of QT using Fridericia's Correction Formula (QTcF) ≥ 500 msec, or at high risk for QT/QTc prolongation.
10. Evidence of hepatic dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2025-11-18 (Actual); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | Treatment Day 42
  To compare all-cause mortality (ACM) at Day 42 following treatment with olorofim versus treatment with AmBisome® followed by standard of care (SOC) in the intent-to-treat (ITT) population of patients with Invasive Fungal Disease (IFD) caused by proven Invasive Aspergillosis (IA) at any site or probable lower respiratory tract disease (LRTD) Aspergillus species (invasive aspergillosis, IA).

SECONDARY OUTCOMES:
Adjudicated Assessment of Overall outcome | Day 42, Day 84, and End of Treatment (anytime during the study between first administration and Day 84)
  To compare the effects of treatment with olorofim versus treatment with AmBisome® followed by SOC on Data Review Committee (DRC)-adjudicated assessment of overall outcome in patients with proven IA or probable LRTD IA at Day 42, Day 84, and End of Treatment.
Investigator-assessed overall response | Day 14, Day 28, Day 42, Day 84, EOT (End of Treatment - Maximum Treatment 84 days [± 7 Days]), and 4-week Follow-up (FU).
  Investigator-assessed overall response (integrating clinical, radiological, and mycological response).
To compare the effects of treatment with olorofim versus treatment with AmBisome® followed by SOC on Galactomannan index. | Day 14, Day 28, Day 42, Day 84, EOT (End of Treatment - Maximum Treatment 84 days [± 7 Days]) and 4-week Follow-up (FU)
  The Sponsor's expert advisors suggested that an appropriate rule would be a failure of the GM to decline from baseline. The experts also state that they have seen very significant variation on retesting of both BAL and serum GM samples and believe it is more appropriate to state a fixed reduction of ≥ 1.0 units than any percentage reduction.
  These rules are used for changes in GM that document failure of therapy:
  1. Serum: After 8 or more days of treatment, serum GM has neither (1) fallen by ≥ 1 unit nor (2) to < 0.5 based on measurements taken at least 8 days apart.
  2. BAL: After 8 or more days of treatment, positive GM from BAL in a patient with a previous BAL test that did not meet the definition of positive (too low or entirely negative) without regard for the interval of time between samples.
To collect additional olorofim and the disproportionate metabolite H26C pharmacokinetic (PK) data for inclusion in a Population PK model | Day 10, Day 14, Day 21, Day 28, Day 42, Day 56, Day 70, Day 84, and at EOT (End of Treatment - Maximum Treatment 84 days [± 7 Days])
  To collect plasma concentration of olorofim and H26C metabolic for for PK analysis (pre-dose and intensive PK). No non-compartmental PK analysis will be performed on the data relating to pre-dose samples and intensive PK samples, apart from data collected from selected regions, which will be reported separately. All relevant olorofim data will be provided to support population PK modelling, which will be reported separately.
Data Review Committee's Assessment of Patient Mortality | Day 42 and 84 and EOT (End of Treatment - Maximum Treatment 84 days [± 7 Days])
  Study data will be independently assessed by a blinded DRC consisting of independent experts in the diagnosis and management of IA, providing an independent adjudication of each patient's mortality based on the survival status collect at time frame.
Diagnosis of a secondary fungal infection | at any time through End Of Treatment
  To compare incidence of a secondary fungal infection when patients treated with olorofim versus treatment with AmBisome followed by SOC.
Quality of life as measured by the 5 Level 5 Dimension (EQ-5D-5L) at Baseline | Days 14 and EOT (End of Treatment - Maximum Treatment 84 days [± 7 Days])
  To assess patient's quality of life measured by the 5-Level 5-Dimension EuroQol Group Health-related Quality of Life Questionnaire (EQ-5D-5L) in both treatment groups
Survival status | Day 42, Day 84, and End Of Treatment and at the 4 weeks ± 7 days FU
  All-cause mortality will be assessed using survival status at time frame.
Safety Assessment | up to the Day 84 and 4-week Follow-up (FU)
  To monitor incidence of Adverse Events and Serious Adverse Events in both treatment arms (Olorofim or AmBisome followed by Standard of Care).

CONTACTS AND LOCATIONS:
Overall Officials: Johan Maertens, MD, Principal Investigator — UZ Leuven
Locations (140):
- United States (24):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - University of California Davis Health System, Sacramento, California
  - UCSF Helen Diller Medical Center at Parnassus Heights, San Francisco, California
  - University of Florida, Gainesville, Florida
  - Augusta University, Augusta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - NIH Clinical Center ,NIAID,NIH, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Clairvoyant Research Group, LLC, Las Vegas, Nevada
  - Rutgers RWJMS, New Brunswick, New Jersey
  - Weill Cornell Medicine NY Presbyterian Hospital, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke Department of Medicine Infectious Diseases Division, Durham, North Carolina
  - OU Health OU Medical Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Medical Center Health System, Pittsburgh, Pennsylvania
  - Houston Methodist, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Australia (5):
  - Royal NorthShore Hospital, Saint Leonards, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Belgium (4):
  - AZ Sint-Jan, Bruges
  - Hôpital Erasme, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
- Brazil (8):
  - Hospital Felício Rocho, Belo Horizonte, Minas Gerais
  - Santa Casa de Misericórdia de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Santa Casa de Misericórdia de Passos, Passos, Minas Gerais
  - Hospital Erasto Gaertner - Liga Paranaense de Combate ao Câncer, Curitiba, Paraná
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital da Universidade Federal de Santa Maria CEP/UFSM, Santa Maria, Rio Grande do Sul
- Canada (4):
  - University of Alberta Hospital, Edmonton, Alberta
  - Hamilton Health Sciences - Juravinski Site, Hamilton, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario
- China (23):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Institute of Hematology and Blood Diseases Hospital, Xiaobailou, Tianjin Municipality
  - The 1st Affiliated Hosp of Wenzhou Medical University, Wenzhou, Zhejiang
  - Peking University People's Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Xiangya Hospital, Central South University, Changsha
  - Chenzhou No.1 People's Hospital, Chenzhou
  - Fujian Medical University Union Hospital, Fuzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - Nanfang Hospital of Southern Medical University, Guangzhou
  - The First Affiliated Hospital of Zhejiang University school of medicine, Hangzhou
  - Anhui Provincial Hospital, Hefei
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning
  - Shengjing Hospital of China Medical University, Shengyang
  - The Second Hospital of Hebei Medical University, Shijiazhuang
  - Xi'an International Medical Center, Xi'an
  - Henan Provincial People's Hospital, Zhengzhou
- France (9):
  - Institut de Cancérologie de Strasbourg Europe - ICANS, Strasbourg, Bas Rhin
  - CHU Besançon - Hôpital Jean Minjoz, Besançon, Doubs
  - CHU de Besancon, Besançon, Doubs
  - CHU Bordeaux Hopital Saint André, Bordeaux, Gironde
  - Institut Universitaire du Cancer de Toulouse- IUCT-O, Toulouse, Haute Garonne
  - CHU de Rennes - Hôpital Pontchaillou, Rennes, Ille-et-Vilaine
  - CHU de Nantes CIC Hematologie, Nantes, Loire Atlantique
  - Hospital Claude Huriez, Lille, Nord
  - Hôpital Necker - Enfants Malades, Paris, Paris
- Germany (4):
  - Universitatsklinikum Leipzig, Leipzig, Saxony
  - Charite Universitatsmedizin Berlin, Berlin
  - Universitaetsklinikum Koeln, Cologne
  - UKE Universitaetsklinikum-Hamburg Eppendorf, Hamburg-Eppendorf
- Israel (4):
  - Soroka University Medical Center, Beersheba
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center Pt, Tel Aviv
- Italy (11):
  - Azienda Ospedaliera Universitaria Luigi Vanvitelli, Napoli, Campania
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, Di Monza E Della Brianza
  - Istituto Clinico Humanitas, Rozzano, Milano
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Ospedale San Raffaele, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - AOU Policlinico di Modena, Modena
  - Clinica Malattie Infettive Dipartimento di Medicina e Chirurgia dell'Università, Perugia
  - Azienda Ospedaliero Universitaria Pisana (Presidio di Cisanello), Pisa
  - Inmi Lazzaro Spallanzani Irccs, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
- Japan (13):
  - Chiba University Hospital, Chiba, Chiba
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Tohoku University Hospital, Sendai, Miyagi
  - Osaka International Cancer Institute, Osaka, Osaka
  - Osaka Metropolitan University Hospital, Osaka, Osaka
  - Kindai University Hospital, Ōsaka-sayama, Osaka
  - The Jikei University Hospital, Minato-Ku, Tokyo
  - Toranomon Hospital, Minatoku, Tokyo to
  - Tokyo Metropolitan Cancer and Infectious diseases Center Komagome Hospital, Bunkyō City
  - Nagasaki University Hospital, Nagasaki
  - Okayama University Hospital, Okayama
  - Saitama Medical Center Jichi Medical University, Saitama
  - Jichi Medical University Hospital, Shimotsuke
- Netherlands (2):
  - Radboud Nijmegen, Nijmegen
  - UMC Utrecht, Utrecht
- New Zealand (2):
  - Wellington Regional Hospital, Newtown, Wellington Region
  - Auckland City Hospital, Auckland
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore General Hospital- Parent, Singapore
- South Korea (2):
  - The Catholic University of Korea, Bucheon-si, Seoul
  - Samsung Medical Center, Irwon-dong, Seoul
- Spain (7):
  - Hospital General Universitario Gregorio Marañón, Retiro, Madrid
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
- Taiwan (5):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taipei Medical University - Shuang Ho Hospital, Ministry of Health and Welfare, New Taipei City
  - China Medical University Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
  - National Taiwan University Hospital, Taipei
- Thailand (2):
  - Siriraj Hospital, Bangkok Noi, Bangkok
  - Srinagarind Hospital, Khon Kaen
- Turkey (Türkiye) (6):
  - Hacettepe University Medical Faculty, Ankara
  - Ankara City Hospital, Ankara
  - Dicle University, Medical Faculty, Diyarbakır
  - Acibadem Atakent Hospital, Istanbul
  - Ege University Medical Faculty, Izmir
  - Ondokuz Mayis Univ. Med. Fac., Samsun
- United Kingdom (3):
  - University Hospital of Wales, Cardiff, Wales
  - Kings College Hospital, London
  - Imperial College London, London